CLINICAL TRIAL: NCT05368077
Title: Brain Changes in Pediatric Obstructive Sleep Apnea
Brief Title: Brain Changes in Pediatric OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Rajesh Kumar, PhD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#21-000408
Record Dates: First submitted 2022-04-11; First posted 2022-05-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Obstructive Sleep Apnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 35 Pediatric Obstructive Sleep Apnea (Experimental): The investigators will also determine whether brain tissue changes, reduced CBF, and altered neural responses to cognitive challenge reverse, and cognition and mood signs improve after standard surgical procedure "adenotonsillectomy" for breathing condition at 6 months in pediatric OSA.
  Interventions: Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: Adenotonsillectomy — Adenotonsillectomy is a standard surgical procedure for pediatric OSA treatment, which involves removal of hypertrophied tonsils and adenoids.

SUMMARY:
Obstructive sleep apnea (OSA) is highly prevalent in children and is often caused by overgrowth of the child's adenoids and/or tonsils. Consequently, adenotonsillectomy (removal of the tonsils and adenoids) is the most common treatment of OSA in children, although just the tonsils or adenoids may be removed depending on the case. As well, OSA in children is often associated with cognitive dysfunction and mood issues, suggesting brain changes due to the condition. However, the link between brain changes, cognitive and moods issues, and OSA in children has not been thoroughly explored. Therefore, this study aims to examine brain changes, cognition and mood in pediatric OSA subjects compared to controls as well as before and after removal of the adenoids and/or tonsils. This study hopes to enroll 70 subjects, ages 7-12 years, 35 healthy controls and 35 subjects diagnosed with OSA and scheduled for an adenoidectomy and/or tonsillectomy. Control subjects will schedule one visit to UCLA and OSA subjects will schedule two. Upon the first visit, all subjects will undergo cognitive, mood and sleep questionnaires and MRI scanning. That will be the duration of the controls' participation in the study; however, OSA subjects will return 6 months later (after their adenoidectomy and/ or tonsillectomy) to repeat the same procedures. Sleep quality, mood, cognition and brain images will be compared between OSA and controls and between OSA subjects before surgery and after surgery.

DETAILED DESCRIPTION:
Pediatric obstructive sleep apnea (OSA) is a common and progressive syndrome accompanied by severe cognition, mood, and daytime behavioral issues, as well as poor school performance, presumably stemming from compromised neural tissue, induced by intermittent hypoxia and perfusion changes. However, it is unclear whether the brain tissue injury is in acute or chronic condition, and whether myelin is preferentially affected than axons, an essential step to understand, since interventions for neural repair/recovery differ for acute vs chronic and myelin vs axonal injury. Also, it is unclear whether accompanying brain changes in pediatric OSA have functional consequences, resulting to cognitive or mood deficits. In addition, intermittent hypoxia triggers a cascade of injurious processes affecting endothelial cells, but unclear whether regional cerebral blood flow (CBF) is reduced in pediatric OSA. Treatment methods for pediatric OSA include tonsillectomy and/or adenoidectomy, and it is unclear whether brain tissue changes, regional CBF, and neural responses to cognitive challenge improve post-treatment. Using diffusion tensor imaging (DTI) and diffusion kurtosis imaging (DKI)-based procedures, acute and chronic tissue changes and axonal status and myelin integrity can be assessed. Regional brain CBF can be assessed by validated arterial spin labeling (ASL) imaging, and regional neural activity to cognitive challenge can be examined with blood-oxygen-level-dependent (BOLD) functional magnetic resonance imaging (MRI). Thus, using 35 treatment-naïve, pediatric OSA and 35 control children, the specific aims are to; determine the nature and types of brain tissue injury, using DTI and DKI measures, in untreated pediatric OSA over healthy controls; identify regional brain CBF, using ASL imaging, and neural responses to cognitive challenge, using BOLD functional MRI in pediatric OSA over healthy children; assess cognitive (by the differential ability scale II and NEPSY II) and emotion functions (by the child behavior checklist) in pediatric OSA compared to control children, and examine relationships between brain injury and cognitive and emotion dysfunctions in pediatric OSA; and examine whether brain tissue changes, reduced CBF, and altered neural responses to cognitive challenge reverse, and cognition and mood signs improve after adenotonsillectomy at 6 months in pediatric OSA. In summary, the nature and types of brain injury, regional CBF changes, and neural responses to cognitive challenge, and whether brain tissue changes, altered CBF, and diminished neural responses, as well as mood and cognitive functions recover after adenotonsillectomy in pediatric OSA will be examined. Evaluation of pathological characteristics is essential to assess the mechanisms of damage, and to suggest intervention strategies before and after surgery. The findings will also help guide potential treatments to rescue/restore brain tissue (e.g., nonsteroidal anti-inflammatory drugs) and improve CBF that could be implemented to benefit cognitive and mood health, and improve academic performance in pediatric OSA.

ELIGIBILITY:
Inclusion Criteria:

OSA

* Pediatric OSA subjects will be in the age range 7-12 years (upper and lower age limit will be chosen to avoid developmental-related brain changes and potential requirement of anesthesia for brain MRI)
* Have a diagnosis of at least moderate OSA (AHI>5 events/hour) via overnight polysomnography at a sleep laboratory
* Without obesity (≥95th percentile BMI for age and sex) to avoid perioperative issues
* No treatment for the breathing condition
* Undergoing for adenotonsillectomy.

Control subjects

* Healthy children
* Age-range from 7-12 years (within ±3 months)
* Sex- and BMI-matched (±2 kg/m2) to pediatric OSA
* No medications for brain disorders
* Without any diagnosed neurological condition

Exclusion Criteria:

* Previous history of diagnosed psychiatric diseases (depression and other brain disorders that may introduce brain injury)
* Cystic fibrosis, concussion, and presence of space-occupying brain lesions
* Metallic or electronic implants and other MRI-specific exclusion criteria

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Brain tissue changes between baseline and after adenotonsillectomy. | 6 months
  The investigators will examine whether brain tissue changes reverse after adenotonsillectomy in pediatric obstructive sleep apnea subjects. The investigators will use diffusion tensor imaging based mean diffusivity and diffusion kurtosis imaging based mean kurtosis measures to examine brain tissue changes; both procedures examine brain tissue integrity with mean diffusivity showing reduced and mean kurtosis indicating increased values in acute tissue changes, and with mean diffusivity showing increased and mean kurtosis showing reduced values in chronic tissue changes.
Regional brain cerebral blood flow changes between baseline and after adenotonsillectomy. | 6 months
  Using arterial spin labeling magnetic resonance imaging, the investigators will assess if regional cerebral blood flow improves after standard obstructive sleep apnea surgery in pediatric subjects. The cerebral blood flow values reduce with hypo-perfusion and increase with hyper-perfusion.
Neural response changes before and after adenotonsillectomy. | 6 months
  Using functional magnetic resonance imaging, the investigators will examine whether neural responses in brain cognitive control sites to arithmetic cognitive challenge will improve after adenotonsillectomy compared to baseline in pediatric obstructive sleep apnea subjects.
Cognitive symptoms examination after adenotonsillectomy surgery. | 6 months
  The investigators will examine cognitive symptom changes after adenotonsillectomy in pediatric obstructive sleep apnea subjects. The investigators will use the Differential Ability Scale II for cognition evaluation. The Differential Ability Scale II scores range from 30-170, with reduced values indicating impaired cognition (General Conceptual Ability score <90, abnormal; General Conceptual Ability score > 90-170, normal).
Cognition assessment after adenotonsillectomy in pediatric obstructive sleep apnea patients. | 6 months
  The investigators will assess cognition changes after adenotonsillectomy in pediatric obstructive sleep apnea subjects. The investigators will use the NEuroPSYchological Assessment II for cognition examination. The NEuroPSYchological Assessment II scores will be lower with impaired cognition (Scaled score <8, abnormal; Scaled score 8-19, normal).
Mood changes after adenotonsillectomy surgery. | 6 months
  The investigators will examine mood changes after adenotonsillectomy in pediatric obstructive sleep apnea subjects using the Child Behavior Checklist. The Child Behavior Checklist scores will be higher with mood symptoms in pediatric obstructive sleep apnea compared to control children (t-scores, 65-69 borderline; >70 clinical).

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the findings have been published, the MRI data (devoid of individual identifiers) will be placed on a read-only anonymous file transfer protocol (ftp) server, with access in the conventional fashion by email ID. Investigators, who request access to the data, will e-mail us with an academic e-mail address and provide a description of their proposed project/purpose. Access to the data will be given to requesting investigator, as long as project does not require personal identifiable information. Such storage represents a substantial commitment of capacity, since the data are expected to require several terabytes. The MRI data (both pre- and post-surgery at 6 months), cognition and mood scores, and OSA disease severity from the same population will be especially valuable to the field, as it is rare to have from patients with pediatric OSA.
Supporting Information: CSR
Time Frame: One year after study completion.

REFERENCES:
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Redline S, Amin R, Beebe D, Chervin RD, Garetz SL, Giordani B, Marcus CL, Moore RH, Rosen CL, Arens R, Gozal D, Katz ES, Mitchell RB, Muzumdar H, Taylor HG, Thomas N, Ellenberg S. The Childhood Adenotonsillectomy Trial (CHAT): rationale, design, and challenges of a randomized controlled trial evaluating a standard surgical procedure in a pediatric population. Sleep. 2011 Nov 1;34(11):1509-17. doi: 10.5665/sleep.1388. PMID 22043122
- [Background] Redline S, Tishler PV, Schluchter M, Aylor J, Clark K, Graham G. Risk factors for sleep-disordered breathing in children. Associations with obesity, race, and respiratory problems. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1527-32. doi: 10.1164/ajrccm.159.5.9809079. PMID 10228121
- [Background] Rosen CL, Larkin EK, Kirchner HL, Emancipator JL, Bivins SF, Surovec SA, Martin RJ, Redline S. Prevalence and risk factors for sleep-disordered breathing in 8- to 11-year-old children: association with race and prematurity. J Pediatr. 2003 Apr;142(4):383-9. doi: 10.1067/mpd.2003.28. PMID 12712055
- [Background] Kumar R, Chavez AS, Macey PM, Woo MA, Yan-Go FL, Harper RM. Altered global and regional brain mean diffusivity in patients with obstructive sleep apnea. J Neurosci Res. 2012 Oct;90(10):2043-52. doi: 10.1002/jnr.23083. Epub 2012 Jun 20. PMID 22715089
- [Background] Kumar R, Pham TT, Macey PM, Woo MA, Yan-Go FL, Harper RM. Abnormal myelin and axonal integrity in recently diagnosed patients with obstructive sleep apnea. Sleep. 2014 Apr 1;37(4):723-32. doi: 10.5665/sleep.3578. PMID 24899761
- [Background] Tummala S, Palomares J, Kang DW, Park B, Woo MA, Harper RM, Kumar R. Global and Regional Brain Non-Gaussian Diffusion Changes in Newly Diagnosed Patients with Obstructive Sleep Apnea. Sleep. 2016 Jan 1;39(1):51-7. doi: 10.5665/sleep.5316. PMID 26285005
- [Background] Tummala S, Roy B, Vig R, Park B, Kang DW, Woo MA, Aysola R, Harper RM, Kumar R. Non-Gaussian Diffusion Imaging Shows Brain Myelin and Axonal Changes in Obstructive Sleep Apnea. J Comput Assist Tomogr. 2017 Mar/Apr;41(2):181-189. doi: 10.1097/RCT.0000000000000537. PMID 27801694
- [Background] Canessa N, Castronovo V, Cappa SF, Aloia MS, Marelli S, Falini A, Alemanno F, Ferini-Strambi L. Obstructive sleep apnea: brain structural changes and neurocognitive function before and after treatment. Am J Respir Crit Care Med. 2011 May 15;183(10):1419-26. doi: 10.1164/rccm.201005-0693OC. Epub 2010 Oct 29. PMID 21037021
- [Background] Castronovo V, Scifo P, Castellano A, Aloia MS, Iadanza A, Marelli S, Cappa SF, Strambi LF, Falini A. White matter integrity in obstructive sleep apnea before and after treatment. Sleep. 2014 Sep 1;37(9):1465-75. doi: 10.5665/sleep.3994. PMID 25142557
- [Background] Ehlert, L., Roy, B., Sahib, A., Song, X., Singh, S., Townsley, M., Kang, D.W., Aysola, R., Wen, E., Woo, M.A., Harper, R.M. & Kumar, R. Diffusion tensor imaging shows brain tissue changes before and after positive airway pressure treatment in patients with obstructive sleep apnea. Society for Neuroscience Annual Meeting, Washington, DC, USA, 2017.
- [Background] Maresky HS, Shpirer I, Klar MM, Levitt M, Sasson E, Tal S. Continuous positive airway pressure alters brain microstructure and perfusion patterns in patients with obstructive sleep apnea. Sleep Med. 2019 May;57:61-69. doi: 10.1016/j.sleep.2018.12.027. Epub 2019 Jan 31. PMID 30897457
- [Background] Rosenzweig I, Glasser M, Crum WR, Kempton MJ, Milosevic M, McMillan A, Leschziner GD, Kumari V, Goadsby P, Simonds AK, Williams SC, Morrell MJ. Changes in Neurocognitive Architecture in Patients with Obstructive Sleep Apnea Treated with Continuous Positive Airway Pressure. EBioMedicine. 2016 May;7:221-9. doi: 10.1016/j.ebiom.2016.03.020. Epub 2016 Mar 25. PMID 27322475
- [Background] Sahib, A., Roy, B., Song, X., Singh, S., Aysola, R., Kang, D.W., Woo, M.A. & Kumar, R. Brain axonal and myelin changes after positive airway pressure treatment in patients with obstructive sleep apnea. Joint Annual Meeting International Society for Magnetic Resonance in Medicine, Paris, France, 2018.
- [Background] Chen HL, Lin HC, Lu CH, Chen PC, Huang CC, Chou KH, Su MC, Friedman M, Chen YW, Lin WC. Systemic inflammation and alterations to cerebral blood flow in obstructive sleep apnea. J Sleep Res. 2017 Dec;26(6):789-798. doi: 10.1111/jsr.12553. Epub 2017 May 17. PMID 28513057
- [Background] Joo EY, Tae WS, Han SJ, Cho JW, Hong SB. Reduced cerebral blood flow during wakefulness in obstructive sleep apnea-hypopnea syndrome. Sleep. 2007 Nov;30(11):1515-20. doi: 10.1093/sleep/30.11.1515. PMID 18041484
- [Background] Yadav SK, Kumar R, Macey PM, Richardson HL, Wang DJ, Woo MA, Harper RM. Regional cerebral blood flow alterations in obstructive sleep apnea. Neurosci Lett. 2013 Oct 25;555:159-64. doi: 10.1016/j.neulet.2013.09.033. Epub 2013 Sep 26. PMID 24076138
- [Background] Lumeng JC, Chervin RD. Epidemiology of pediatric obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):242-52. doi: 10.1513/pats.200708-135MG. PMID 18250218
- [Background] Barone JG, Hanson C, DaJusta DG, Gioia K, England SJ, Schneider D. Nocturnal enuresis and overweight are associated with obstructive sleep apnea. Pediatrics. 2009 Jul;124(1):e53-9. doi: 10.1542/peds.2008-2805. PMID 19564269
- [Background] Nieminen P, Lopponen T, Tolonen U, Lanning P, Knip M, Lopponen H. Growth and biochemical markers of growth in children with snoring and obstructive sleep apnea. Pediatrics. 2002 Apr;109(4):e55. doi: 10.1542/peds.109.4.e55. PMID 11927728
- [Background] Suratt PM, Barth JT, Diamond R, D'Andrea L, Nikova M, Perriello VA Jr, Carskadon MA, Rembold C. Reduced time in bed and obstructive sleep-disordered breathing in children are associated with cognitive impairment. Pediatrics. 2007 Feb;119(2):320-9. doi: 10.1542/peds.2006-1969. PMID 17272622
- [Background] Soultan Z, Wadowski S, Rao M, Kravath RE. Effect of treating obstructive sleep apnea by tonsillectomy and/or adenoidectomy on obesity in children. Arch Pediatr Adolesc Med. 1999 Jan;153(1):33-7. doi: 10.1001/archpedi.153.1.33. PMID 9894997
- [Background] Series F, Cormier Y, La Forge J. [Physiopathology of obstructive sleep apneas]. Rev Mal Respir. 1989;6(5):397-407. French. PMID 2690208
- [Background] Gozal D, Wang M, Pope DW Jr. Objective sleepiness measures in pediatric obstructive sleep apnea. Pediatrics. 2001 Sep;108(3):693-7. doi: 10.1542/peds.108.3.693. PMID 11533338
- [Background] Beebe DW, Ris MD, Kramer ME, Long E, Amin R. The association between sleep disordered breathing, academic grades, and cognitive and behavioral functioning among overweight subjects during middle to late childhood. Sleep. 2010 Nov;33(11):1447-56. doi: 10.1093/sleep/33.11.1447. PMID 21102986
- [Background] Crabtree VM, Varni JW, Gozal D. Health-related quality of life and depressive symptoms in children with suspected sleep-disordered breathing. Sleep. 2004 Sep 15;27(6):1131-8. doi: 10.1093/sleep/27.6.1131. PMID 15532207
- [Background] Gozal D. Sleep-disordered breathing and school performance in children. Pediatrics. 1998 Sep;102(3 Pt 1):616-20. doi: 10.1542/peds.102.3.616. PMID 9738185
- [Background] Kheirandish L, Gozal D. Neurocognitive dysfunction in children with sleep disorders. Dev Sci. 2006 Jul;9(4):388-99. doi: 10.1111/j.1467-7687.2006.00504.x. PMID 16764612
- [Background] O'Brien LM, Mervis CB, Holbrook CR, Bruner JL, Smith NH, McNally N, McClimment MC, Gozal D. Neurobehavioral correlates of sleep-disordered breathing in children. J Sleep Res. 2004 Jun;13(2):165-72. doi: 10.1111/j.1365-2869.2004.00395.x. PMID 15175097
- [Background] Cha J, Zea-Hernandez JA, Sin S, Graw-Panzer K, Shifteh K, Isasi CR, Wagshul ME, Moran EE, Posner J, Zimmerman ME, Arens R. The Effects of Obstructive Sleep Apnea Syndrome on the Dentate Gyrus and Learning and Memory in Children. J Neurosci. 2017 Apr 19;37(16):4280-4288. doi: 10.1523/JNEUROSCI.3583-16.2017. Epub 2017 Mar 20. PMID 28320844
- [Background] Halbower AC, Degaonkar M, Barker PB, Earley CJ, Marcus CL, Smith PL, Prahme MC, Mahone EM. Childhood obstructive sleep apnea associates with neuropsychological deficits and neuronal brain injury. PLoS Med. 2006 Aug;3(8):e301. doi: 10.1371/journal.pmed.0030301. PMID 16933960
- [Background] Horne RSC, Roy B, Walter LM, Biggs SN, Tamanyan K, Weichard A, Nixon GM, Davey MJ, Ditchfield M, Harper RM, Kumar R. Regional brain tissue changes and associations with disease severity in children with sleep-disordered breathing. Sleep. 2018 Feb 1;41(2):zsx203. doi: 10.1093/sleep/zsx203. PMID 29267958
- [Background] Kheirandish-Gozal L, Sahib AK, Macey PM, Philby MF, Gozal D, Kumar R. Regional brain tissue integrity in pediatric obstructive sleep apnea. Neurosci Lett. 2018 Aug 24;682:118-123. doi: 10.1016/j.neulet.2018.06.002. Epub 2018 Jun 5. PMID 29883682
- [Background] Kheirandish-Gozal L, Yoder K, Kulkarni R, Gozal D, Decety J. Preliminary functional MRI neural correlates of executive functioning and empathy in children with obstructive sleep apnea. Sleep. 2014 Mar 1;37(3):587-92. doi: 10.5665/sleep.3504. PMID 24587582
- [Background] Macey PM, Kheirandish-Gozal L, Prasad JP, Ma RA, Kumar R, Philby MF, Gozal D. Altered Regional Brain Cortical Thickness in Pediatric Obstructive Sleep Apnea. Front Neurol. 2018 Jan 22;9:4. doi: 10.3389/fneur.2018.00004. eCollection 2018. PMID 29403430
- [Background] Philby MF, Macey PM, Ma RA, Kumar R, Gozal D, Kheirandish-Gozal L. Reduced Regional Grey Matter Volumes in Pediatric Obstructive Sleep Apnea. Sci Rep. 2017 Mar 17;7:44566. doi: 10.1038/srep44566. PMID 28303917
- [Background] Chopra S, Polotsky VY, Jun JC. Sleep Apnea Research in Animals. Past, Present, and Future. Am J Respir Cell Mol Biol. 2016 Mar;54(3):299-305. doi: 10.1165/rcmb.2015-0218TR. PMID 26448201
- [Background] Gozal D, Row BW, Gozal E, Kheirandish L, Neville JJ, Brittian KR, Sachleben LR Jr, Guo SZ. Temporal aspects of spatial task performance during intermittent hypoxia in the rat: evidence for neurogenesis. Eur J Neurosci. 2003 Oct;18(8):2335-42. doi: 10.1046/j.1460-9568.2003.02947.x. PMID 14622195
- [Background] Gozal E, Row BW, Schurr A, Gozal D. Developmental differences in cortical and hippocampal vulnerability to intermittent hypoxia in the rat. Neurosci Lett. 2001 Jun 15;305(3):197-201. doi: 10.1016/s0304-3940(01)01853-5. PMID 11403939
- [Background] Xu W, Chi L, Row BW, Xu R, Ke Y, Xu B, Luo C, Kheirandish L, Gozal D, Liu R. Increased oxidative stress is associated with chronic intermittent hypoxia-mediated brain cortical neuronal cell apoptosis in a mouse model of sleep apnea. Neuroscience. 2004;126(2):313-23. doi: 10.1016/j.neuroscience.2004.03.055. PMID 15207349
- [Background] Huang YS, Guilleminault C, Lee LA, Lin CH, Hwang FM. Treatment outcomes of adenotonsillectomy for children with obstructive sleep apnea: a prospective longitudinal study. Sleep. 2014 Jan 1;37(1):71-6. doi: 10.5665/sleep.3310. PMID 24470697
- [Background] Basser PJ, Mattiello J, LeBihan D. Estimation of the effective self-diffusion tensor from the NMR spin echo. J Magn Reson B. 1994 Mar;103(3):247-54. doi: 10.1006/jmrb.1994.1037. PMID 8019776
- [Background] Pierpaoli C, Jezzard P, Basser PJ, Barnett A, Di Chiro G. Diffusion tensor MR imaging of the human brain. Radiology. 1996 Dec;201(3):637-48. doi: 10.1148/radiology.201.3.8939209.
- [Background] Jensen JH, Falangola MF, Hu C, Tabesh A, Rapalino O, Lo C, Helpern JA. Preliminary observations of increased diffusional kurtosis in human brain following recent cerebral infarction. NMR Biomed. 2011 Jun;24(5):452-7. doi: 10.1002/nbm.1610. Epub 2010 Oct 19. PMID 20960579
- [Background] Cheung MM, Hui ES, Chan KC, Helpern JA, Qi L, Wu EX. Does diffusion kurtosis imaging lead to better neural tissue characterization? A rodent brain maturation study. Neuroimage. 2009 Apr 1;45(2):386-92. doi: 10.1016/j.neuroimage.2008.12.018. Epub 2008 Dec 25. PMID 19150655
- [Background] Hui ES, Cheung MM, Qi L, Wu EX. Towards better MR characterization of neural tissues using directional diffusion kurtosis analysis. Neuroimage. 2008 Aug 1;42(1):122-34. doi: 10.1016/j.neuroimage.2008.04.237. Epub 2008 Apr 30. PMID 18524628
- [Background] Mori S, Zhang J. Principles of diffusion tensor imaging and its applications to basic neuroscience research. Neuron. 2006 Sep 7;51(5):527-39. doi: 10.1016/j.neuron.2006.08.012. PMID 16950152
- [Background] Nair G, Tanahashi Y, Low HP, Billings-Gagliardi S, Schwartz WJ, Duong TQ. Myelination and long diffusion times alter diffusion-tensor-imaging contrast in myelin-deficient shiverer mice. Neuroimage. 2005 Oct 15;28(1):165-74. doi: 10.1016/j.neuroimage.2005.05.049. Epub 2005 Jul 14. PMID 16023870
- [Background] Song SK, Sun SW, Ramsbottom MJ, Chang C, Russell J, Cross AH. Dysmyelination revealed through MRI as increased radial (but unchanged axial) diffusion of water. Neuroimage. 2002 Nov;17(3):1429-36. doi: 10.1006/nimg.2002.1267. PMID 12414282
- [Background] Trip SA, Wheeler-Kingshott C, Jones SJ, Li WY, Barker GJ, Thompson AJ, Plant GT, Miller DH. Optic nerve diffusion tensor imaging in optic neuritis. Neuroimage. 2006 Apr 1;30(2):498-505. doi: 10.1016/j.neuroimage.2005.09.024. Epub 2005 Oct 20. PMID 16242968
- [Background] de Bazelaire C, Alsop DC, George D, Pedrosa I, Wang Y, Michaelson MD, Rofsky NM. Magnetic resonance imaging-measured blood flow change after antiangiogenic therapy with PTK787/ZK 222584 correlates with clinical outcome in metastatic renal cell carcinoma. Clin Cancer Res. 2008 Sep 1;14(17):5548-54. doi: 10.1158/1078-0432.CCR-08-0417. PMID 18765547
- [Background] Hu WT, Wang Z, Lee VM, Trojanowski JQ, Detre JA, Grossman M. Distinct cerebral perfusion patterns in FTLD and AD. Neurology. 2010 Sep 7;75(10):881-8. doi: 10.1212/WNL.0b013e3181f11e35. PMID 20819999
- [Background] Feng CM, Narayana S, Lancaster JL, Jerabek PA, Arnow TL, Zhu F, Tan LH, Fox PT, Gao JH. CBF changes during brain activation: fMRI vs. PET. Neuroimage. 2004 May;22(1):443-6. doi: 10.1016/j.neuroimage.2004.01.017. PMID 15110037
- [Background] Ye FQ, Berman KF, Ellmore T, Esposito G, van Horn JD, Yang Y, Duyn J, Smith AM, Frank JA, Weinberger DR, McLaughlin AC. H(2)(15)O PET validation of steady-state arterial spin tagging cerebral blood flow measurements in humans. Magn Reson Med. 2000 Sep;44(3):450-6. doi: 10.1002/1522-2594(200009)44:33.0.co;2-0. PMID 10975898
- [Background] Chen Y, Wang DJ, Detre JA. Test-retest reliability of arterial spin labeling with common labeling strategies. J Magn Reson Imaging. 2011 Apr;33(4):940-9. doi: 10.1002/jmri.22345. PMID 21448961
- [Background] Floyd TF, Ratcliffe SJ, Wang J, Resch B, Detre JA. Precision of the CASL-perfusion MRI technique for the measurement of cerebral blood flow in whole brain and vascular territories. J Magn Reson Imaging. 2003 Dec;18(6):649-55. doi: 10.1002/jmri.10416. PMID 14635149
- [Background] Wang J, Aguirre GK, Kimberg DY, Roc AC, Li L, Detre JA. Arterial spin labeling perfusion fMRI with very low task frequency. Magn Reson Med. 2003 May;49(5):796-802. doi: 10.1002/mrm.10437. PMID 12704760
- [Background] Canivez GL, McGill RJ. Factor structure of the Differential Ability Scales-Second Edition: Exploratory and hierarchical factor analyses with the core subtests. Psychol Assess. 2016 Nov;28(11):1475-1488. doi: 10.1037/pas0000279. Epub 2016 Jan 25. PMID 27046278
- [Background] Keith, T.Z., Low, J.A., Reynolds, M.R., Patel, P.G. & Ridley, K.P. Higher-order factor structure of the differential ability scales-II: consistency across ages 4 to 17. Psychology in the Schools 47: 676-697, 2010.
- [Background] Achenbach, T.M. The child behavior checklist and related instruments. In: The use of psychological testing for treatment planning and outcomes assessment, 2nd ed, edited by. Mahwah, NJ, US: Lawrence Erlbaum Associates Publishers, 1999, p. 429-466.
- [Background] Achenbach TM, Ruffle TM. The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies. Pediatr Rev. 2000 Aug;21(8):265-71. doi: 10.1542/pir.21-8-265. No abstract available. PMID 10922023
- [Background] Ellis, E.M., Zarndt, R., Ho, B., Hopkins, S. & Powell, F.L. Effects of non-steroid anti-inflammatory drugs on the human hypoxic ventilatory response and acclimatization. The FASEB Journal 26: 1150.1152- 1150.1152, 2012.
- [Background] Goswami AR, Dutta G, Ghosh T. Naproxen, a Nonsteroidal Anti-Inflammatory Drug, Can Affect Daily Hypobaric Hypoxia-Induced Alterations of Monoamine Levels in Different Areas of the Brain in Male Rats. High Alt Med Biol. 2016 Jun;17(2):133-40. doi: 10.1089/ham.2015.0052. Epub 2016 Feb 19. PMID 26894935
- [Background] Ishiguro H, Kawahara T. Nonsteroidal anti-inflammatory drugs and prostatic diseases. Biomed Res Int. 2014;2014:436123. doi: 10.1155/2014/436123. Epub 2014 May 12. PMID 24900965
- [Background] Daniel DG, Weinberger DR, Jones DW, Zigun JR, Coppola R, Handel S, Bigelow LB, Goldberg TE, Berman KF, Kleinman JE. The effect of amphetamine on regional cerebral blood flow during cognitive activation in schizophrenia. J Neurosci. 1991 Jul;11(7):1907-17. doi: 10.1523/JNEUROSCI.11-07-01907.1991. PMID 2066768
- [Background] Dormehl IC, Jordaan B, Oliver DW, Croft S. SPECT monitoring of improved cerebral blood flow during long-term treatment of elderly patients with nootropic drugs. Clin Nucl Med. 1999 Jan;24(1):29-34. doi: 10.1097/00003072-199901000-00007. PMID 9890490
- [Background] Lipsitz LA, Gagnon M, Vyas M, Iloputaife I, Kiely DK, Sorond F, Serrador J, Cheng DM, Babikian V, Cupples LA. Antihypertensive therapy increases cerebral blood flow and carotid distensibility in hypertensive elderly subjects. Hypertension. 2005 Feb;45(2):216-21. doi: 10.1161/01.HYP.0000153094.09615.11. Epub 2005 Jan 17. PMID 15655124
- [Background] Serrador JM, Freeman R. Enhanced Cholinergic Activity Improves Cerebral Blood Flow during Orthostatic Stress. Front Neurol. 2017 Mar 20;8:103. doi: 10.3389/fneur.2017.00103. eCollection 2017. PMID 28373858
- [Background] Warwick JP, Mason DG. Obstructive sleep apnoea syndrome in children. Anaesthesia. 1998 Jun;53(6):571-9. doi: 10.1046/j.1365-2044.1998.00370.x. PMID 9709144
- [Background] Kheirandish-Gozal L, De Jong MR, Spruyt K, Chamuleau SA, Gozal D. Obstructive sleep apnoea is associated with impaired pictorial memory task acquisition and retention in children. Eur Respir J. 2010 Jul;36(1):164-9. doi: 10.1183/09031936.00114209. Epub 2010 Jan 14. PMID 20075057
- [Background] Tan HL, Gozal D, Kheirandish-Gozal L. Obstructive sleep apnea in children: a critical update. Nat Sci Sleep. 2013 Sep 25;5:109-23. doi: 10.2147/NSS.S51907. PMID 24109201
- [Background] Bass JL, Corwin M, Gozal D, Moore C, Nishida H, Parker S, Schonwald A, Wilker RE, Stehle S, Kinane TB. The effect of chronic or intermittent hypoxia on cognition in childhood: a review of the evidence. Pediatrics. 2004 Sep;114(3):805-16. doi: 10.1542/peds.2004-0227. PMID 15342857
- [Background] Blunden SL, Beebe DW. The contribution of intermittent hypoxia, sleep debt and sleep disruption to daytime performance deficits in children: consideration of respiratory and non-respiratory sleep disorders. Sleep Med Rev. 2006 Apr;10(2):109-18. doi: 10.1016/j.smrv.2005.11.003. Epub 2006 Feb 20. PMID 16488632
- [Background] Urschitz MS, Guenther A, Eggebrecht E, Wolff J, Urschitz-Duprat PM, Schlaud M, Poets CF. Snoring, intermittent hypoxia and academic performance in primary school children. Am J Respir Crit Care Med. 2003 Aug 15;168(4):464-8. doi: 10.1164/rccm.200212-1397OC. Epub 2003 May 28. PMID 12773324
- [Background] Trosman I, Trosman SJ. Cognitive and Behavioral Consequences of Sleep Disordered Breathing in Children. Med Sci (Basel). 2017 Dec 1;5(4):30. doi: 10.3390/medsci5040030. PMID 29194375
- [Background] Bedard MA, Montplaisir J, Richer F, Rouleau I, Malo J. Obstructive sleep apnea syndrome: pathogenesis of neuropsychological deficits. J Clin Exp Neuropsychol. 1991 Nov;13(6):950-64. doi: 10.1080/01688639108405110. PMID 1779033
- [Background] Engleman H, Joffe D. Neuropsychological function in obstructive sleep apnoea. Sleep Med Rev. 1999 Mar;3(1):59-78. doi: 10.1016/s1087-0792(99)90014-x. PMID 15310490
- [Background] Owens J, Spirito A, Marcotte A, McGuinn M, Berkelhammer L. Neuropsychological and Behavioral Correlates of Obstructive Sleep Apnea Syndrome in Children: A Preliminary Study. Sleep Breath. 2000;4(2):67-78. doi: 10.1007/BF03045026. PMID 11868122
- [Background] Zhao J, Han S, Zhang J, Wang G, Wang H, Xu Z, Tai J, Peng X, Guo Y, Liu H, Tian J, Jin X, Zheng L, Zhang J, Ni X. Association between mild or moderate obstructive sleep apnea-hypopnea syndrome and cognitive dysfunction in children. Sleep Med. 2018 Oct;50:132-136. doi: 10.1016/j.sleep.2018.04.009. Epub 2018 Jun 9. PMID 30036785
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Friedman BC, Hendeles-Amitai A, Kozminsky E, Leiberman A, Friger M, Tarasiuk A, Tal A. Adenotonsillectomy improves neurocognitive function in children with obstructive sleep apnea syndrome. Sleep. 2003 Dec 15;26(8):999-1005. doi: 10.1093/sleep/26.8.999. PMID 14746381
- [Background] Goldstein NA, Post JC, Rosenfeld RM, Campbell TF. Impact of tonsillectomy and adenoidectomy on child behavior. Arch Otolaryngol Head Neck Surg. 2000 Apr;126(4):494-8. doi: 10.1001/archotol.126.4.494. PMID 10772303
- [Background] Marcus CL, Moore RH, Rosen CL, Giordani B, Garetz SL, Taylor HG, Mitchell RB, Amin R, Katz ES, Arens R, Paruthi S, Muzumdar H, Gozal D, Thomas NH, Ware J, Beebe D, Snyder K, Elden L, Sprecher RC, Willging P, Jones D, Bent JP, Hoban T, Chervin RD, Ellenberg SS, Redline S; Childhood Adenotonsillectomy Trial (CHAT). A randomized trial of adenotonsillectomy for childhood sleep apnea. N Engl J Med. 2013 Jun 20;368(25):2366-76. doi: 10.1056/NEJMoa1215881. Epub 2013 May 21. PMID 23692173
- [Background] Murata E, Mohri I, Kato-Nishimura K, Iimura J, Ogawa M, Tachibana M, Ohno Y, Taniike M. Evaluation of behavioral change after adenotonsillectomy for obstructive sleep apnea in children with autism spectrum disorder. Res Dev Disabil. 2017 Jun;65:127-139. doi: 10.1016/j.ridd.2017.04.012. Epub 2017 May 14. PMID 28514706
- [Background] Taylor HG, Bowen SR, Beebe DW, Hodges E, Amin R, Arens R, Chervin RD, Garetz SL, Katz ES, Moore RH, Morales KH, Muzumdar H, Paruthi S, Rosen CL, Sadhwani A, Thomas NH, Ware J, Marcus CL, Ellenberg SS, Redline S, Giordani B. Cognitive Effects of Adenotonsillectomy for Obstructive Sleep Apnea. Pediatrics. 2016 Aug;138(2):e20154458. doi: 10.1542/peds.2015-4458. PMID 27464674
- [Background] Torretta S, Rosazza C, Pace ME, Iofrida E, Marchisio P. Impact of adenotonsillectomy on pediatric quality of life: review of the literature. Ital J Pediatr. 2017 Nov 25;43(1):107. doi: 10.1186/s13052-017-0424-2. PMID 29178907
- [Background] Gozal D, Daniel JM, Dohanich GP. Behavioral and anatomical correlates of chronic episodic hypoxia during sleep in the rat. J Neurosci. 2001 Apr 1;21(7):2442-50. doi: 10.1523/JNEUROSCI.21-07-02442.2001. PMID 11264318
- [Background] Pae EK, Chien P, Harper RM. Intermittent hypoxia damages cerebellar cortex and deep nuclei. Neurosci Lett. 2005 Feb 28;375(2):123-8. doi: 10.1016/j.neulet.2004.10.091. Epub 2004 Dec 2. PMID 15670654
- [Background] Veasey SC, Davis CW, Fenik P, Zhan G, Hsu YJ, Pratico D, Gow A. Long-term intermittent hypoxia in mice: protracted hypersomnolence with oxidative injury to sleep-wake brain regions. Sleep. 2004 Mar 15;27(2):194-201. doi: 10.1093/sleep/27.2.194. PMID 15124711
- [Background] Zhang JH, Fung SJ, Xi M, Sampogna S, Chase MH. Apnea produces neuronal degeneration in the pons and medulla of guinea pigs. Neurobiol Dis. 2010 Oct;40(1):251-64. doi: 10.1016/j.nbd.2010.05.032. Epub 2010 Jun 8. PMID 20554036
- [Background] Dirnagl U, Iadecola C, Moskowitz MA. Pathobiology of ischaemic stroke: an integrated view. Trends Neurosci. 1999 Sep;22(9):391-7. doi: 10.1016/s0166-2236(99)01401-0. PMID 10441299
- [Background] Hossmann KA. Cortical steady potential, impedance and excitability changes during and after total ischemia of cat brain. Exp Neurol. 1971 Aug;32(2):163-75. doi: 10.1016/0014-4886(71)90060-4. No abstract available. PMID 5567067
- [Background] LOWRY OH, PASSONNEAU JV, HASSELBERGER FX, SCHULZ DW. EFFECT OF ISCHEMIA ON KNOWN SUBSTRATES AND COFACTORS OF THE GLYCOLYTIC PATHWAY IN BRAIN. J Biol Chem. 1964 Jan;239:18-30. No abstract available. PMID 14114842
- [Background] O'Dell TJ, Huang PL, Dawson TM, Dinerman JL, Snyder SH, Kandel ER, Fishman MC. Endothelial NOS and the blockade of LTP by NOS inhibitors in mice lacking neuronal NOS. Science. 1994 Jul 22;265(5171):542-6. doi: 10.1126/science.7518615.
- [Background] Oehmichen M, Ochs U, Meissner C. Regional potassium distribution in the brain in forensic relevant types of intoxication preliminary morphometric evaluation using a histochemical method. Neurotoxicology. 2001 Feb;22(1):99-107. doi: 10.1016/s0161-813x(00)00005-x. PMID 11307856
- [Background] Mintorovitch J, Yang GY, Shimizu H, Kucharczyk J, Chan PH, Weinstein PR. Diffusion-weighted magnetic resonance imaging of acute focal cerebral ischemia: comparison of signal intensity with changes in brain water and Na+,K(+)-ATPase activity. J Cereb Blood Flow Metab. 1994 Mar;14(2):332-6. doi: 10.1038/jcbfm.1994.40. PMID 8113328
- [Background] Benveniste H, Drejer J, Schousboe A, Diemer NH. Elevation of the extracellular concentrations of glutamate and aspartate in rat hippocampus during transient cerebral ischemia monitored by intracerebral microdialysis. J Neurochem. 1984 Nov;43(5):1369-74. doi: 10.1111/j.1471-4159.1984.tb05396.x. PMID 6149259
- [Background] Hagberg H, Lehmann A, Sandberg M, Nystrom B, Jacobson I, Hamberger A. Ischemia-induced shift of inhibitory and excitatory amino acids from intra- to extracellular compartments. J Cereb Blood Flow Metab. 1985 Sep;5(3):413-9. doi: 10.1038/jcbfm.1985.56. PMID 4030918
- [Background] Kassmann CM, Nave KA. Oligodendroglial impact on axonal function and survival - a hypothesis. Curr Opin Neurol. 2008 Jun;21(3):235-41. doi: 10.1097/WCO.0b013e328300c71f. PMID 18451704
- [Background] Nukada H, Dyck PJ. Acute ischemia causes axonal stasis, swelling, attenuation, and secondary demyelination. Ann Neurol. 1987 Sep;22(3):311-8. doi: 10.1002/ana.410220306. PMID 3674796
- [Background] Shereen A, Nemkul N, Yang D, Adhami F, Dunn RS, Hazen ML, Nakafuku M, Ning G, Lindquist DM, Kuan CY. Ex vivo diffusion tensor imaging and neuropathological correlation in a murine model of hypoxia-ischemia-induced thrombotic stroke. J Cereb Blood Flow Metab. 2011 Apr;31(4):1155-69. doi: 10.1038/jcbfm.2010.212. Epub 2010 Dec 8. PMID 21139628
- [Background] Matsumoto K, Lo EH, Pierce AR, Wei H, Garrido L, Kowall NW. Role of vasogenic edema and tissue cavitation in ischemic evolution on diffusion-weighted imaging: comparison with multiparameter MR and immunohistochemistry. AJNR Am J Neuroradiol. 1995 May;16(5):1107-15. PMID 7639135
- [Background] Kidwell CS, Alger JR, Di Salle F, Starkman S, Villablanca P, Bentson J, Saver JL. Diffusion MRI in patients with transient ischemic attacks. Stroke. 1999 Jun;30(6):1174-80. doi: 10.1161/01.str.30.6.1174. PMID 10356095
- [Background] Lecouvet FE, Duprez TP, Raymackers JM, Peeters A, Cosnard G. Resolution of early diffusion-weighted and FLAIR MRI abnormalities in a patient with TIA. Neurology. 1999 Mar 23;52(5):1085-7. doi: 10.1212/wnl.52.5.1085. PMID 10102438
- [Background] Basser PJ, Pierpaoli C. Microstructural and physiological features of tissues elucidated by quantitative-diffusion-tensor MRI. J Magn Reson B. 1996 Jun;111(3):209-19. doi: 10.1006/jmrb.1996.0086. PMID 8661285
- [Background] Basser PJ, Mattiello J, LeBihan D. MR diffusion tensor spectroscopy and imaging. Biophys J. 1994 Jan;66(1):259-67. doi: 10.1016/S0006-3495(94)80775-1. PMID 8130344
- [Background] Le Bihan D, Mangin JF, Poupon C, Clark CA, Pappata S, Molko N, Chabriat H. Diffusion tensor imaging: concepts and applications. J Magn Reson Imaging. 2001 Apr;13(4):534-46. doi: 10.1002/jmri.1076. PMID 11276097
- [Background] Basser PJ, Pierpaoli C. A simplified method to measure the diffusion tensor from seven MR images. Magn Reson Med. 1998 Jun;39(6):928-34. doi: 10.1002/mrm.1910390610. PMID 9621916
- [Background] Ahlhelm F, Schneider G, Backens M, Reith W, Hagen T. Time course of the apparent diffusion coefficient after cerebral infarction. Eur Radiol. 2002 Sep;12(9):2322-9. doi: 10.1007/s00330-001-1291-0. Epub 2002 Mar 19. PMID 12195489
- [Background] Hossmann KA, Fischer M, Bockhorst K, Hoehn-Berlage M. NMR imaging of the apparent diffusion coefficient (ADC) for the evaluation of metabolic suppression and recovery after prolonged cerebral ischemia. J Cereb Blood Flow Metab. 1994 Sep;14(5):723-31. doi: 10.1038/jcbfm.1994.93. PMID 8063868
- [Background] Loubinoux I, Volk A, Borredon J, Guirimand S, Tiffon B, Seylaz J, Meric P. Spreading of vasogenic edema and cytotoxic edema assessed by quantitative diffusion and T2 magnetic resonance imaging. Stroke. 1997 Feb;28(2):419-26; discussion 426-7. doi: 10.1161/01.str.28.2.419. PMID 9040700
- [Background] Chan KC, Khong PL, Lau HF, Cheung PT, Wu EX. Late measures of microstructural alterations in severe neonatal hypoxic-ischemic encephalopathy by MR diffusion tensor imaging. Int J Dev Neurosci. 2009 Oct;27(6):607-15. doi: 10.1016/j.ijdevneu.2009.05.012. Epub 2009 Jun 6. PMID 19505567
- [Background] Kelly PJ, Hedley-Whyte ET, Primavera J, He J, Gonzalez RG. Diffusion MRI in ischemic stroke compared to pathologically verified infarction. Neurology. 2001 Apr 10;56(7):914-20. doi: 10.1212/wnl.56.7.914. PMID 11294929
- [Background] Warach S, Mosley M, Sorensen AG, Koroshetz W. Time course of diffusion imaging abnormalities in human stroke. Stroke. 1996 Jul;27(7):1254-6. No abstract available. PMID 8685940
- [Background] Newcombe VF, Williams GB, Nortje J, Bradley PG, Harding SG, Smielewski P, Coles JP, Maiya B, Gillard JH, Hutchinson PJ, Pickard JD, Carpenter TA, Menon DK. Analysis of acute traumatic axonal injury using diffusion tensor imaging. Br J Neurosurg. 2007 Aug;21(4):340-8. doi: 10.1080/02688690701400882. PMID 17676452
- [Background] Bhagat YA, Hussain MS, Stobbe RW, Butcher KS, Emery DJ, Shuaib A, Siddiqui MM, Maheshwari P, Al-Hussain F, Beaulieu C. Elevations of diffusion anisotropy are associated with hyper-acute stroke: a serial imaging study. Magn Reson Imaging. 2008 Jun;26(5):683-93. doi: 10.1016/j.mri.2008.01.015. Epub 2008 Apr 28. PMID 18440747
- [Background] Yang Q, Tress BM, Barber PA, Desmond PM, Darby DG, Gerraty RP, Li T, Davis SM. Serial study of apparent diffusion coefficient and anisotropy in patients with acute stroke. Stroke. 1999 Nov;30(11):2382-90. doi: 10.1161/01.str.30.11.2382. PMID 10548675
- [Background] Counsell SJ, Shen Y, Boardman JP, Larkman DJ, Kapellou O, Ward P, Allsop JM, Cowan FM, Hajnal JV, Edwards AD, Rutherford MA. Axial and radial diffusivity in preterm infants who have diffuse white matter changes on magnetic resonance imaging at term-equivalent age. Pediatrics. 2006 Feb;117(2):376-86. doi: 10.1542/peds.2005-0820. PMID 16452356
- [Background] Lowe MJ, Horenstein C, Hirsch JG, Marrie RA, Stone L, Bhattacharyya PK, Gass A, Phillips MD. Functional pathway-defined MRI diffusion measures reveal increased transverse diffusivity of water in multiple sclerosis. Neuroimage. 2006 Sep;32(3):1127-33. doi: 10.1016/j.neuroimage.2006.04.208. Epub 2006 Jun 23. PMID 16798013
- [Background] Pierpaoli C, Barnett A, Pajevic S, Chen R, Penix LR, Virta A, Basser P. Water diffusion changes in Wallerian degeneration and their dependence on white matter architecture. Neuroimage. 2001 Jun;13(6 Pt 1):1174-85. doi: 10.1006/nimg.2001.0765. PMID 11352623
- [Background] Jensen JH, Helpern JA, Ramani A, Lu H, Kaczynski K. Diffusional kurtosis imaging: the quantification of non-gaussian water diffusion by means of magnetic resonance imaging. Magn Reson Med. 2005 Jun;53(6):1432-40. doi: 10.1002/mrm.20508. PMID 15906300
- [Background] Lu H, Jensen JH, Ramani A, Helpern JA. Three-dimensional characterization of non-gaussian water diffusion in humans using diffusion kurtosis imaging. NMR Biomed. 2006 Apr;19(2):236-47. doi: 10.1002/nbm.1020. PMID 16521095
- [Background] Tabesh A, Jensen JH, Ardekani BA, Helpern JA. Estimation of tensors and tensor-derived measures in diffusional kurtosis imaging. Magn Reson Med. 2011 Mar;65(3):823-36. doi: 10.1002/mrm.22655. Epub 2010 Oct 28. PMID 21337412
- [Background] Fieremans E, Jensen JH, Helpern JA. White matter characterization with diffusional kurtosis imaging. Neuroimage. 2011 Sep 1;58(1):177-88. doi: 10.1016/j.neuroimage.2011.06.006. Epub 2011 Jun 13. PMID 21699989
- [Background] Lazar M, Jensen JH, Xuan L, Helpern JA. Estimation of the orientation distribution function from diffusional kurtosis imaging. Magn Reson Med. 2008 Oct;60(4):774-81. doi: 10.1002/mrm.21725. PMID 18816827
- [Background] Wang DJ, Chen Y, Fernandez-Seara MA, Detre JA. Potentials and challenges for arterial spin labeling in pharmacological magnetic resonance imaging. J Pharmacol Exp Ther. 2011 May;337(2):359-66. doi: 10.1124/jpet.110.172577. Epub 2011 Feb 11. PMID 21317356
- [Background] Buckley DL, Bui JD, Phillips MI, Zelles T, Inglis BA, Plant HD, Blackband SJ. The effect of ouabain on water diffusion in the rat hippocampal slice measured by high resolution NMR imaging. Magn Reson Med. 1999 Jan;41(1):137-42. doi: 10.1002/(sici)1522-2594(199901)41:13.0.co;2-y. PMID 10025621
- [Background] Mulkern RV, Zengingonul HP, Robertson RL, Bogner P, Zou KH, Gudbjartsson H, Guttmann CR, Holtzman D, Kyriakos W, Jolesz FA, Maier SE. Multi-component apparent diffusion coefficients in human brain: relationship to spin-lattice relaxation. Magn Reson Med. 2000 Aug;44(2):292-300. doi: 10.1002/1522-2594(200008)44:23.0.co;2-q. PMID 10918329
- [Background] Vestergaard-Poulsen P, Hansen B, Ostergaard L, Jakobsen R. Microstructural changes in ischemic cortical gray matter predicted by a model of diffusion-weighted MRI. J Magn Reson Imaging. 2007 Sep;26(3):529-40. doi: 10.1002/jmri.21030. PMID 17685422
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Goodwin JL, Vasquez MM, Silva GE, Quan SF. Incidence and remission of sleep-disordered breathing and related symptoms in 6- to 17-year old children--the Tucson Children's Assessment of Sleep Apnea Study. J Pediatr. 2010 Jul;157(1):57-61. doi: 10.1016/j.jpeds.2010.01.033. Epub 2010 Mar 20. PMID 20304429
- [Background] Li AM, So HK, Au CT, Ho C, Lau J, Ng SK, Abdullah VJ, Fok TF, Wing YK. Epidemiology of obstructive sleep apnoea syndrome in Chinese children: a two-phase community study. Thorax. 2010 Nov;65(11):991-7. doi: 10.1136/thx.2010.134858. PMID 20965935
- [Background] Ehlert, L., Roy, B., Sahib, A.K., Song, X., Singh, S., Townsley, M., Kang, D.W., Aysola, R., Wen, E., Woo, M.A., Harper, R.M. & Kumar, R. Diffusion tensor imaging shows brain tissue changes before and after positive airway pressure treatment in patients with obstructive sleep apnea. Society for Neuroscience Annual Meeting, Washington, D.C., 2017.
- [Background] Kim H, Joo E, Suh S, Kim JH, Kim ST, Hong SB. Effects of long-term treatment on brain volume in patients with obstructive sleep apnea syndrome. Hum Brain Mapp. 2016 Jan;37(1):395-409. doi: 10.1002/hbm.23038. Epub 2015 Oct 27. PMID 26503297
- [Background] Kumar R, Delshad S, Macey PM, Woo MA, Harper RM. Development of T2-relaxation values in regional brain sites during adolescence. Magn Reson Imaging. 2011 Feb;29(2):185-93. doi: 10.1016/j.mri.2010.08.006. Epub 2010 Oct 8. PMID 20933351
- [Background] Kumar R, Delshad S, Woo MA, Macey PM, Harper RM. Age-related regional brain T2-relaxation changes in healthy adults. J Magn Reson Imaging. 2012 Feb;35(2):300-8. doi: 10.1002/jmri.22831. Epub 2011 Oct 10. PMID 21987489
- [Background] Kumar R, Macey PM, Woo MA, Alger JR, Harper RM. Diffusion tensor imaging demonstrates brainstem and cerebellar abnormalities in congenital central hypoventilation syndrome. Pediatr Res. 2008 Sep;64(3):275-80. doi: 10.1203/PDR.0b013e31817da10a. PMID 18458651
- [Background] Kumar R, Macey PM, Woo MA, Alger JR, Harper RM. Elevated mean diffusivity in widespread brain regions in congenital central hypoventilation syndrome. J Magn Reson Imaging. 2006 Dec;24(6):1252-8. doi: 10.1002/jmri.20759. PMID 17075838
- [Background] Kumar R, Macey PM, Woo MA, Alger JR, Keens TG, Harper RM. Neuroanatomic deficits in congenital central hypoventilation syndrome. J Comp Neurol. 2005 Jul 11;487(4):361-71. doi: 10.1002/cne.20565. PMID 15906312
- [Background] Kumar R, Nguyen HD, Macey PM, Woo MA, Harper RM. Dilated basilar arteries in patients with congenital central hypoventilation syndrome. Neurosci Lett. 2009 Dec 25;467(2):139-43. doi: 10.1016/j.neulet.2009.10.024. Epub 2009 Oct 12. PMID 19822189
- [Background] Kumar R, Nguyen HD, Macey PM, Woo MA, Harper RM. Regional brain axial and radial diffusivity changes during development. J Neurosci Res. 2012 Feb;90(2):346-55. doi: 10.1002/jnr.22757. Epub 2011 Sep 21. PMID 21938736
- [Background] Macey PM, Alger JR, Kumar R, Macey KE, Woo MA, Harper RM. Global BOLD MRI changes to ventilatory challenges in congenital central hypoventilation syndrome. Respir Physiol Neurobiol. 2003 Dec 16;139(1):41-50. doi: 10.1016/j.resp.2003.09.006. PMID 14637309
- [Background] American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):268-86. doi: 10.1097/ALN.0000000000000053. No abstract available. PMID 24346178
- [Background] Dehlink E, Tan HL. Update on paediatric obstructive sleep apnoea. J Thorac Dis. 2016 Feb;8(2):224-35. doi: 10.3978/j.issn.2072-1439.2015.12.04. PMID 26904263
- [Background] Paruthi, S. Evaluation of suspected obstructive sleep apnea in children. Edited by A.G. Hoppin, 2019.
- [Background] Rubinstein, B.J. & Baldassari, C.M. An Update on the management of pediatric obstructive sleep apnea. Curr Treat Options Pediatr 1: 211-223, 2015.
- [Background] Wolfe RM, Pomerantz J, Miller DE, Weiss-Coleman R, Solomonides T. Obstructive Sleep Apnea: Preoperative Screening and Postoperative Care. J Am Board Fam Med. 2016 Mar-Apr;29(2):263-75. doi: 10.3122/jabfm.2016.02.150085. PMID 26957384
- [Background] Elliott, C.D. Differential Ability Scales : introductory and technical handbook. San Antonio: Psychological Corp: Harcourt Brace Jovanovich, 1990.
- [Background] Achenbach TM, R.L. Manual for the ASEBA school-based forms and profiles. Burlington: University of Vermont, Research Center for Children , Youth and Families, 2001.
- [Background] Barmpoutis, A. & Jiachen, Z. Diffusion kurtosis imaging: robust estimation from DW-MRI using homogeneous polynomials. 2011 IEEE International Symposium on Biomedical Imaging: From Nano to Macro, Chicago, IL: 262-265, 2011.
- [Background] Barmpoutis A, Vemuri BC. A UNIFIED FRAMEWORK FOR ESTIMATING DIFFUSION TENSORS OF ANY ORDER WITH SYMMETRIC POSITIVE-DEFINITE CONSTRAINTS. Proc IEEE Int Symp Biomed Imaging. 2010 Apr 14:1385-1388. doi: 10.1109/ISBI.2010.5490256. PMID 21594011
- [Background] Ashburner J, Friston KJ. Unified segmentation. Neuroimage. 2005 Jul 1;26(3):839-51. doi: 10.1016/j.neuroimage.2005.02.018. Epub 2005 Apr 1. PMID 15955494
- [Background] Woo MA, Palomares JA, Macey PM, Fonarow GC, Harper RM, Kumar R. Global and regional brain mean diffusivity changes in patients with heart failure. J Neurosci Res. 2015 Apr;93(4):678-85. doi: 10.1002/jnr.23525. Epub 2014 Dec 13. PMID 25502071
- [Background] Wang J, Zhang Y, Wolf RL, Roc AC, Alsop DC, Detre JA. Amplitude-modulated continuous arterial spin-labeling 3.0-T perfusion MR imaging with a single coil: feasibility study. Radiology. 2005 Apr;235(1):218-28. doi: 10.1148/radiol.2351031663. Epub 2005 Feb 16. PMID 15716390
- [Background] Ogren JA, Macey PM, Kumar R, Woo MA, Harper RM. Central autonomic regulation in congenital central hypoventilation syndrome. Neuroscience. 2010 Jun 2;167(4):1249-56. doi: 10.1016/j.neuroscience.2010.02.078. Epub 2010 Mar 6. PMID 20211704
- [Background] Chumbley JR, Friston KJ. False discovery rate revisited: FDR and topological inference using Gaussian random fields. Neuroimage. 2009 Jan 1;44(1):62-70. doi: 10.1016/j.neuroimage.2008.05.021. Epub 2008 May 23. PMID 18603449
- [Background] Bender HA, Marks BC, Brown ER, Zach L, Zaroff CM. Neuropsychologic performance of children with epilepsy on the NEPSY. Pediatr Neurol. 2007 May;36(5):312-7. doi: 10.1016/j.pediatrneurol.2007.01.011. PMID 17509463
- [Background] Leviton A, Joseph RM, Allred EN, O'Shea TM, Taylor HG, Kuban KKC. Antenatal and Neonatal Antecedents of Executive Dysfunctions in Extremely Preterm Children. J Child Neurol. 2018 Mar;33(3):198-208. doi: 10.1177/0883073817750499. Epub 2018 Jan 11. PMID 29322860
- [Background] Lind A, Korkman M, Lehtonen L, Lapinleimu H, Parkkola R, Matomaki J, Haataja L; PIPARI Study Group. Cognitive and neuropsychological outcomes at 5 years of age in preterm children born in the 2000s. Dev Med Child Neurol. 2011 Mar;53(3):256-62. doi: 10.1111/j.1469-8749.2010.03828.x. Epub 2010 Dec 17. PMID 21166668
- [Background] Spencer-Smith MM, Spittle AJ, Lee KJ, Doyle LW, Anderson PJ. Bayley-III Cognitive and Language Scales in Preterm Children. Pediatrics. 2015 May;135(5):e1258-65. doi: 10.1542/peds.2014-3039. Epub 2015 Apr 20. PMID 25896835

DOCUMENTS (1):
  • Informed Consent Form (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT05368077/ICF_000.pdf